CLINICAL TRIAL: NCT07166133
Title: GORE® TAG® Thoracic Branch Endoprosthesis Zone 0/1 Post-Approval Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBE 25-03
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Aortic Arch Dissection; Aortic Arch Aneurysm
Keywords: Zone 0; Zone 1
MeSH Terms: conditions — Dissection, Thoracic Aorta; Aneurysm, Aortic Arch

STUDY DESIGN:
Intervention Model Description: GORE® TAG® Thoracic Branch Endoprosthesis (TBE)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- GORE® TAG® Thoracic Branch Endoprosthesis (TBE Device) (Other)
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® TAG® Thoracic Branch Endoprosthesis — Lesions in aortic arch in Zone 0 or Zone 1

SUMMARY:
A prospective multi-center post-market study collecting outcomes through at least 5-years and up to 10-years post procedure for subjects treated with the TBE Device in Zone 0/1 as part of routine clinical practice.

DETAILED DESCRIPTION:
Minimum of 125 total subjects with a TBE Device implantation procedure initiated in up to 50 Sites in the United States. Subjects will have follow-up at 1 Month, 6 Month, 1 Year, and annually thereafter for a minimum of 5-years and up to a maximum of 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative (LAR) provides written authorization and/or consent per institution and geographical requirements.
2. Patient has been or is intended to be treated with the TBE Device in Zone 0 or Zone 1.
3. Patient is age ≥ 18 years at time of informed consent signature.

Exclusion Criteria:

1. Patient who is, at the time of consent, unlikely to be available for defined follow-up visits.
2. Patient with exclusion criteria required by local law.
3. Patient is currently enrolled in or plans to enroll in any concurrent investigational drug and/or investigational device study within 12 months of study enrollment. Subjects cannot be enrolled in another Gore study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with index endovascular procedure initiated after (or following) the surgical revascularization procedure | Index Endovascular Procedure Only
  Great vessel surgical revascularization procedure is completed, and the endovascular implantation procedure is initiated for the implantation of the TBE Device, without interim death or study discontinuation.
Device Technical Success (index procedure only) | Index Endovascular Procedure Only
  * Successful access, delivery, and accurate deployment of the device to the intended location, and retrieval of the delivery system.
  * Patency of the endovascular aortic and side branch components.
  * The absence of any unanticipated additional corrective procedure related to the device, procedure, or withdrawal of the delivery system.
Lesion-related mortality | Within 30 days of surgical revascularization or within 30 days of index endovascular procedure
  Death meeting at least one of the following characteristics:
  * Death during the hospitalization or within 30 days following the surgical revascularization procedure.
  * Death during the hospitalization or within 30 days following the index endovascular procedure or following conversion to open repair.
  * Death during the hospitalization or within 30 days following a complication from a secondary procedure associated with the index lesion or study device.
  * Any death where the treated disease / index lesion or study device caused or significantly contributed to the death, including lesion-rupture, aortic-related complications, disease progression involving the index lesion.
Disabling Stroke | Within 30 days of surgical revascularization or within 30 days of index endovascular procedure
  Stroke is the acute onset of symptoms consistent with focal or multifocal central nervous system (CNS) injury caused by vascular blockage resulting in ischemia or vascular rupture resulting in hemorrhage, that:
  * Is identified within 30-days following the surgical revascularization procedure or within 30-days following the index endovascular procedure -AND-
  * Persists for ≥ 24 hours or until death, or has symptoms lasting < 24 hours, with pathology or neuroimaging confirmation of CNS infarction -AND-
  * Has an mRS ≥ 2 with an increase from baseline of at least one grade due to neurological deficits at no more than 120 days post index endovascular procedure.
Permanent Paraplegia (within 30-days) | Within 30 days of index endovascular procedure
  Paraplegia secondary to Spinal Cord Ischemia identified within 30 days following the index endovascular procedure combined with Spinal Cord Ischemia scale grade = 3 at the one-month follow-up visit. Paraplegia will be assessed using the SVS spinal cord ischemia grading system
Permanent Paraparesis (within 30-days) | Within 30 days of index endovascular procedure
  Paraparesis secondary to Spinal Cord Ischemia identified within 30 days following the index endovascular procedure, combined with Spinal Cord Ischemia scale grade = 2 at the one-month follow-up visit. Paraparesis will be assessed using the SVS spinal cord ischemia grading system.
New onset renal failure (within 30-days) requiring on-going dialysis | Within 30 days of index endovascular procedure
  New onset of sustained renal failure identified within 30 days following the index endovascular procedure, combined with requiring dialysis at the 1-Month follow-up visit.
Lesion rupture (treated area) | Minimum of 60 months and up to a maximum 120 months
  Rupture in the treated segment of the vessel (e.g., aorta or branch) verified with direct observation or CT / CTA scan.
Loss of aortic or branch patency | Minimum of 60 months and up to a maximum of 120 months
  No flow or contrast detected through the implanted aortic component or endovascular branch component confirmed with imaging and/or direct observation.
Endoleaks | Minimum of 60 months and up to a maximum of 120 months
  Perfusion of a treated lesion via:
  * Type I endoleak is defined as a sealing failure at one of the attachment zones of the graft to the vessel wall, whereby arterial flow perfuses the treated lesion via a perigraft channel:
    * Type Ia: Proximal aortic attachment zone
    * Type Ib: Distal aortic attachment zone
    * Type Ic: Distal attachment zone for branch component.
  * Type II: Retrograde flow from native aortic branch arteries.
  * Type III endoleak: Component disconnection or fabric disruption resulting in arterial flow into the perigraft space:
    * Type IIIa: Attachment of aortic components (aortic-aortic)
    * Type IIIb: Fabric tear or disruption
    * Type IIIc: Attachment of aortic component-side-branch or side-branch-side-branch.
  * Type IV: Late endoleak due to flow through porous fabric.
  * Type V/Endotension: Aneurysm sac enlargement > 5 mm with no imaging evidence of an endoleak.
  * Indeterminate: Endoleak is identified, but source cannot be ascertained.
Reintervention | Minimum of 60 months and up to a maximum of 120 months
  Additional surgical or interventional procedure related to the treated disease / index lesion, the study device, or to the treatment / procedure.
  This may include surgical or interventional treatment for endoleaks, disease progression, procedures on the branch to improve or restore patency, spinal drains for Spinal Cord Injury (SCI) management, or conversion to open surgery.
  Events will not include access site(s) complications, interventions to address issues related to non-treated area of the index lesion, such as bare stent implantation to address bowel ischemia associated with aortic dissection.

SECONDARY OUTCOMES:
Access-related complications (index endovascular procedure only) | Index endovascular procedure only
  Complications associated with the access sites used during treatment and any subsequent unplanned access-related reinterventions. This may include pseudoaneurysm, thrombosis, or complications associated with percutaneous closure devices.
Life threatening bleed (index endovascular procedure only) | Index endovascular procedure only
  An event associated with the index endovascular procedure leading to any of the following events as prior to discharge:
  * Overt bleeding requiring a transfusion of ≥5 units of whole blood/red blood cells within 48 hours of index endovascular procedure.
  * Cardiac tamponade
  * Overt bleeding requiring reoperation, surgical exploration, or reintervention for the purpose of controlling bleeding
  * Bleeding requiring intravenous vasoactive drugs
  * Fatal bleeding is bleeding that directly causes death with no other explainable cause
Stroke | Minimum of 60 months and up to a maximum of 120 months
  Stroke is the acute onset of symptoms consistent with focal or multifocal central nervous system (CNS) injury caused by vascular blockage resulting in ischemia or vascular rupture resulting in hemorrhage, that:
  * Persists for ≥ 24 hours or until death -OR-
  * Symptoms lasting < 24 hours, with pathology or neuroimaging confirmation of CNS infarction.
  Disabling stroke will be determined based on mRS ≥ 2 with an increase from baseline of at least one grade due to neurological deficits at no more than 120 days following the suspected stroke event.
Transient Ischemic Attack (TIA) | Minimum of 60 months and up to a maximum of 120 months
  Transient focal neurological signs or symptoms (lasting < 24 h) presumed to be due to focal brain ischemia but without evidence of acute infarction by neuroimaging or pathology (or in the absence of imaging).
Paraplegia (within 30-days) | Within 30 days of index endovascular procedure
  Paraplegia secondary to Spinal Cord Ischemia identified within 30 days following the index endovascular procedure. Paraplegia will be assessed using the SVS spinal cord ischemia grading system.
Paraparesis (within 30-days) | Within 30 days of index endovascular procedure
  Paraparesis secondary to Spinal Cord Ischemia identified within 30 days following the index endovascular procedure. Paraparesis will be assessed using the SVS spinal cord ischemia grading system.
Distal device-related thromboembolic adverse event requiring intervention or surgery (through 1-Month) | Through 1 Month of index endovascular procedure
  Device-related ischemic events in tissues distal to the device implantation site resulting in bypass, open surgical or transcatheter intervention, limb amputation, or leading to death.
Myocardial infarction (within 30-days) | Within 30 days of surgical revascularization procedure or within 30 days of index endovascular procedure
  Elevated CK-MB (≥ 10x ULN) measured within 48 hours following the surgical revascularization or index endovascular procedure or need for urgent or emergent PCI/CABG within 30-days following the surgical revascularization or index endovascular procedure as confirmed at the 1-Month follow-up visit.
Laryngeal or Phrenic Nerve injury (within 30-days) | Within 30 days of surgical revascularization or within 30 days of index endovascular procedure
  Irreversible laryngeal nerve injury or phrenic nerve injury requiring unplanned surgery or intervention within 30-days following the surgical revascularization or index endovascular procedure as confirmed at the 1-Month follow-up visit.
Fistula formation | Minimum of 60 months and up to a maximum of 120 months
  Fistula detected between the aorta and any adjacent structure associated with the area treated with the endovascular stent graft system verified with direct observation or CT scan.
Upper extremity ischemia | Minimum of 60 months and up to a maximum of 120 months
  Clinically reported, device-related ischemia (Serious Adverse Event) not evident at the time of the index procedure with CTA-verified branch vessel compromise (i.e., malperfusion).
Lesion enlargement (treated area) | Minimum of 60 months and up to maximum of 120 months
  An increase in maximum vessel (e.g., aorta or treated branch) diameter of > 5 mm in the treated region as compared to baseline using orthogonal (i.e., perpendicular to the centerline) measurements on CT / CTA scans
Device migration | Minimum of 60 months and up to a maximum of 120 months
  Longitudinal movement of all or part of the device for a distance ≥ 10 mm, as confirmed by CTA scan, relative to anatomical landmarks and device positioning at the first post-operative CTA scan.
New dissection (with / without treatment) | Minimum of 60 months and up to maximum of 120 months
  A new arterial tear that was not present at the time of initial presentation caused either by a stent graft, natural disease progression or iatrogenic injury during the endovascular procedure. This can include the propagation, or extension, of a previous dissection.
Device integrity events (e.g., fracture, kinking, compression) | Minimum of 60 months and up to maximum of 120 months
  Defined as any of the following:
  * Wire fractures
  * Stent kinking: Narrowing of the stent graft associated with demonstrable angulation in any of the stent components, with demonstrable flow
  * Disruption / tears in the graft component of the stent graft
  * Stent compression or invagination: Transient or permanent stent graft collapse following complete device deployment, resulting in an overall reduction in the vessel luminal diameter
False lumen status (dissection pathology) | Minimum of 60 months and up to maximum of 120 months
  Status of the false lumen both within and outside of the segment of the aorta initially treated with an endovascular stent graft:
  * Patent: Flow present throughout the entire aortic false lumen (absence of thrombus) on arterial-phase or delayed contrast-enhanced imaging.
  * Partial thrombosis: Thrombus or clot within the aortic false lumen but with a residual patent ﬂow channel on arterial-phase or delayed contrast-enhanced imaging.
  * Complete thrombosis: Complete thrombosis of the aortic false lumen on arterial- and delayed-phase imaging.
False lumen perfusion (dissection pathology) | Minimum of 60 months and up to maximum of 120 months
  Flow into the false lumen via:
  * Type IA entry ﬂow: Flow between the proximal endograft and aortic wall allowing systemic pressure antegrade ﬂow into the primary entry tear and proximal false lumen.
  * Type IB entry ﬂow: Distal entry tear adjacent to endograft due to septal fenestration or a new intimal tear at the distal aspect of the stent graft (dSINE) allowing systemic pressure direct ﬂow into the false lumen.
  * Type II entry ﬂow: Retrograde entry ﬂow through arch vessel branches (innominate, carotid, subclavian) or thoracic bronchial and intercostal arteries into the false lumen.
  * Type R entry ﬂow: Antegrade entry ﬂow from the true lumen into the false lumen through distal branch fenestrations (uncovered intercostal arteries, visceral or renal arteries, lumbar arteries, iliac branches) or septal fenestrations (excluding SINE).

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol